CLINICAL TRIAL: NCT03706976
Title: NIRS to Monitor Abdominal Tissue Oxygen Saturation in Preterm Infants in an Open Mono-centric Study
Brief Title: NIRS to Monitor Abdominal Tissue Oxygen Saturation in Preterm Infants
Acronym: CTOM-FIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carag AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2018.7557
Record Dates: First submitted 2018-10-10; First posted 2018-10-16 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Neonatal Disorder
MeSH Terms: conditions — Infant, Newborn, Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CTOM (Experimental)
  Interventions: Device: Tissue Oxygenation Monitoring

INTERVENTIONS:
Device: Tissue Oxygenation Monitoring — The NIRS sensor will be applied to the abdomen of the study population. To ensure good skin contact the sensor will be placed underneath the diaper. If that should not provide enough measurement stability, additional fixation will be given by employing aforementioned flexible bandage routinely employed in neonatal care. Once good skin contact is ensured, the sensor will measure aStO2 for up to seventy-two hours. The presence of this sensor will not disturb daily clinical activities or medical treatment in any way. Should good skin contact be endangered by movements, clinical interactions or such, the sensor will be removed and re-attached to the infants' abdomen as a consequence.

SUMMARY:
The NIRS (near infrared spectroscopy) sensor will be applied to the abdomen of the study population. To ensure good skin contact the sensor will be placed underneath the diaper. If that should not provide enough measurement stability, additional fixation will be given by employing aforementioned flexible bandage routinely employed in neonatal care. Once good skin contact is ensured, the sensor will measure aStO2 (abdominal tissue oxygen saturation) for up to seventy-two hours. The presence of this sensor will not disturb daily clinical activities or medical treatment in any way. Should good skin contact be endangered by movements, clinical interactions or such, the sensor will be removed and re-attached to the infants' abdomen as a consequence.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with GA less than 35 0/7 weeks
* Start of measurement earliest at day of life 2 for preterm infants with GA >=30 0/7 weeks and day of life 4 otherwise. The measurement will not start after day of life 5 for all GA.
* Signed Informed consent of the legal representative(s) is received after being informed. It is sufficient, if the consent form is signed by one legal representative, which is in majority of cases either the mother or the father.
* Clinically stable condition. The clinical stability is to be reconfirmed before the start and checked during the measurement.

Exclusion Criteria:

* Injured, hypersensitive or bruised skin present on the belly,
* Existence of clinical instability at any time during the investigation leads to exclusion, if ordered so by the physician entrusted with the investigation,
* Any medical care equipment, e.g. patches, dressing, umbilical arterial or venous catheter, blood supply, etc., prohibiting correct placement of the sensors,
* Dark skin pigmentation or dense hairiness on the belly absorbing too much light in the near infrared region to allow for NIRS,
* Congenital malformations,
* Severe metabolic disorders,
* Early onset sepsis,
* Inability of legal representatives to understand the purpose of the clinical trial due to language barriers such as the insufficient ability to understand the spoken or written language,
* The treatment of newborn jaundice with light during the intended measurement time,
* Previous enrolment into the current study,
* Family members, employees and other dependent persons of the investigator,
* Participation in another study with investigational drug/device within the preceding days and during the present study which may influence aStO2.

Max Age: 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
Feasibility of aStO2 measurements in all patients | 72 hours
  aStO2 values calculated with and without considering the presence of additional absorbers besides haemoglobin.

SECONDARY OUTCOMES:
Safety of the investigational device assessed by evaluation of adverse events | 72 hours
  Evaluation of AEs (Adverse Event) with regard to the investigational device. The safety related to application and use of the NIRS sensors is aimed for.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsspital Zürich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No